CLINICAL TRIAL: NCT02972528
Title: Allogeneic Defibrinated Platelet Rich Plasma Lysate for the Healing of Chronic Diabetic Foot Ulcer
Brief Title: The Use of Allogenic Platelet Rich Plasma for the Treatment of Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanan Jafar (Other)
Responsible Party: Sponsor-Investigator, Hanan Jafar, Researcher, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFUUJCTC
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU; Diabetic Foot Ulcer; Diabetes; Platelet Rich Plasma
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Lysate (Active Comparator): Patients will receive 5ml peri-lesional injections of Platelet Lysate at weekly intervals, for 4 consecutive times (week 0,1,2,3).
  Interventions: Biological: Platelet Lysate
- Platelet Poor Plasma (Placebo Comparator): Patients will receive 5ml peri-lesional injections of Platelet Poor Plasma at weekly intervals, for 4 consecutive times (week 0,1,2,3).
  Interventions: Biological: Platelet Poor Plasma

INTERVENTIONS:
Biological: Platelet Lysate — Direct injection of allogenic Platelet Lysate
  Arms: Platelet Lysate
Biological: Platelet Poor Plasma — Direct injection of allogenic Platelet Poor Plasma
  Arms: Platelet Poor Plasma

SUMMARY:
Allogenic defibrinated platelet rich plasma lysate will be injected in patients diagnosed with Diabetic Foot Ulcer (DFU).

DETAILED DESCRIPTION:
In this study, allogenic, defibrinated platelet rich plasma lysate will be used as a direct injection into the periphery of diabetic chronic foot ulcers which have not healed using standard of care. Investigators anticipate a significant response in treated individuals measured by the percentage of skin restoration achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with type 1 or type 2 diabetes between the ages of 18 and 70 with an ulcer of at least 4 weeks duration
2. HemoglobinA1C (HbA1c) < 12
3. Index foot ulcer located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces); and wound area (length x width) measurement between 2 cm2 and 20 cm2, inclusive.
4. Wounds located under a Charcot deformity had to be free of acute changes and must have under gone appropriate structural consolidation.
5. The index ulcer had to be clinically non-infected and full - thickness without exposure of bone, ligaments, or tendons.
6. The protocol requires that post debridement the ulcer would be free of necrotic debris, foreign bodies or sinus tracts.
7. Non- invasive vascular testing ankle brachial index (ABI).
8. Physical examination (including a Semmes-Weinstein monofilament test for neuropathy)
9. Blood tests to be obtained Complete Blood Count and HbA1c.
10. Approved, informed, signed consent.
11. Negative test for Hepatitis C (HC), Hepatitis B (HB), Human Immunodeficiency Virus 1 and 2 (HIVI and II), Venereal Disease Research Laboratory (VDRL).

Exclusion Criteria:

1. Patient currently enrolled in another investigational device or drug trial or previously enrolled (within last 30 days) in investigative research of a device or pharmaceutical agent.
2. Ulcer decreased ≥50% in area during 7-day screening period.
3. Ulcer is due to non-diabetic etiology.
4. Patient's blood vessels are non-compressible for ABI testing.
5. Evidence of gangrene in ulcer or on any part of the foot.
6. Patient has radiographic evidence consistent with diagnosis of acute Charcot foot.
7. Patient is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
8. Patient has received growth factor therapy within 7 days of randomization.
9. Screening hemoglobin <10.5 mg/dL.
10. Screening platelet count < 100 x 109/L.
11. Patient is undergoing renal dialysis, has known immune insufficiency, known abnormal platelet activation disorders - ie, gray platelet syndrome, liver disease, active cancer (except remote basal cell of the skin), eating/ nutritional,hematologic, collagen vascular disease, rheumatic disease, or bleeding disorders.
12. History of peripheral vascular repair within the 30 days of randomization
13. Patient has known or suspected osteomyelitis.
14. Surgical correction (other than debridement) required for ulcer to heal.
15. Index ulcer has exposed tendons, ligaments, muscle, or bone.
16. Patient is known to have a psychological, developmental, physical, emotional, or social disorder, or any other situation that may interfere with compliance with study requirements and/or healing of the ulcer
17. History of alcohol or drug abuse within the last year prior to randomization.
18. Patient has inadequate venous access for blood draw.
19. Positive test for HC, HB, HIVI and II, VDRL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-03 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) as a result of the injection | 3 months
  Evaluate the safety of this treatment, by gathering and assessing the number, timing, severity, duration, and resolution of related adverse events.

SECONDARY OUTCOMES:
Assess the efficacy of allogenic Platelet Lysate injection by clinical examination | 4 months
  To determine short term speed and effectiveness of allogeneic, platelet rich plasma lysate on the healing of diabetic foot ulceration compared with Platelet Poor Plasma by measuring the diameter of ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided